CLINICAL TRIAL: NCT00603863
Title: A Phase Ib/II Study of Fractionated 90Y-hPAM4 Plus Gemcitabine in Patients With Previously Untreated Advanced Pancreatic Cancer.
Brief Title: Safety and Efficacy Study of Different Doses of 90Y-hPAM4 Combined With Gemcitabine in Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hPAM4-02
Record Dates: First submitted 2008-01-08; First posted 2008-01-29 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2014-01

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; hPAM4; MUC1 antibody; cancer of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- multiple dose levels (Experimental): 1 of 3 different dose levels of 90Y-hPAM4 given once weekly for 3 weeks along with 4 weekly doses of gemcitabine.
  Interventions: Biological: IMMU-107 (hPAM4)

INTERVENTIONS:
Biological: IMMU-107 (hPAM4) — 90Y-hPAM4 once weekly for 3 weeks gemcitabine once weekly for 4 weeks
  Other Names: hPAM4; IMMU-107; 90Y-hPAM4; anti-mucin antibody

SUMMARY:
This is a study to test whether different doses of 90Y-hPAM4 are safe to give in combination with gemcitabine in patients with previously untreated pancreatic cancer.

DETAILED DESCRIPTION:
Patients receive a 4-week treatment cycle with once-weekly 30-minute gemcitabine infusions beginning one week prior to the first 90Y-hPAM4dose and continuing during the 3 consecutive weeks over which once weekly 90Y-hPAM4 doses are given. Depending on toxicity, patient cohorts will receive one of several possible 90Y and gemcitabine dose combinations. Post-treatment evaluations conducted until instituting another 90YhPAM4 treatment cycle, maintenance gemcitabine or for a maximum period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, >18 years of age, who are able to understand and give written informed consent.
* Histologically or cytologically confirmed pancreatic adenocarcinoma.
* Stage III (locally advanced, unresectable) or Stage IV (metastatic) disease, including patients who underwent surgery but had incomplete resections.
* Treatment naïve (no prior chemotherapy, radiotherapy or investigational agents for pancreatic cancer)
* Karnofsky performance status > 70 % (Appendix A).
* Expected survival > 3 months.
* At least 4 weeks beyond major surgery and recovered from all acute toxicities
* At least 2 weeks beyond corticosteroids, except low doses (i.e., 20 mg/day of prednisone or equivalent) to treat nausea or other illness such as rheumatoid arthritis
* Adequate hematology without ongoing transfusional support (hemoglobin > 11 g/dL, ANC > 2,000 per mm3, platelets > 150,000 per mm3)
* Adequate renal and hepatic function (creatinine and bilirubin ≤ 1.5 X IULN, AST and ALT ≤ 2.0 X IULN)
* Otherwise, all toxicity at study entry <Grade 1 by NCI CTC v3.0.

Exclusion Criteria:

* Women who are pregnant or lactating.

  * Women of childbearing potential and fertile men unwilling to use effective contraception during study until conclusion of 12-week post-treatment evaluation period.
  * Known metastatic disease to the central nervous system.
  * Presence of bulky disease (defined as any single mass >10 cm in its greatest dimension)
  * Patients with >Grade 2 anorexia, nausea or vomiting, and/or signs of intestinal obstruction.
  * Prior radiation dose >3,000 cGy to the liver, >2,000 cGy to lungs and kidneys or prior external beam irradiation to a field that includes more than 30% of the red marrow.
  * Patients with non-melanoma skin cancer or carcinoma in situ of the cervix are not excluded, but patients with other prior malignancies must have had at least a 5-year disease free interval.
  * Patients known to be HIV positive, hepatitis B positive, or hepatitis C positive.
  * Known history of active coronary artery disease, unstable angina, myocardial infarction, or congestive heart failure present within 6 months or cardiac arrhythmia requiring anti-arrhythmia therapy.
  * Known history of active COPD, or other moderate-to-severe respiratory illness present within 6 months.
  * Known autoimmune disease or presence of autoimmune phenomena (except rheumatoid arthritis requiring only low dose maintenance corticosteroids).
  * Infection requiring intravenous antibiotic use within 1 week.
  * Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-01; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
safety will be evaluated based upon physical examinations, hematology and chemistry laboratory testing as well as toxicity | over 12 weeks

SECONDARY OUTCOMES:
Efficacy and Clinical benefit measures such as quality of life, pain assessments, etc. | over 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PHD, Study Chair — Gilead Sciences
Locations (11):
- United States (11):
  - Christiana Care Health Services, Newark, Delaware
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Herbert Werthem College of Medicine/Jackson North Medical Center, Miami, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Winship Cancer Institute/Emory University Hospital, Atlanta, Georgia
  - Goshen Cancer Center, Goshen, Indiana
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Thomas Jefferson University Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Gold DV, Karanjawala Z, Modrak DE, Goldenberg DM, Hruban RH. PAM4-reactive MUC1 is a biomarker for early pancreatic adenocarcinoma. Clin Cancer Res. 2007 Dec 15;13(24):7380-7. doi: 10.1158/1078-0432.CCR-07-1488. PMID 18094420
- [Background] Modrak DE, Gold DV, Goldenberg DM. Sphingolipid targets in cancer therapy. Mol Cancer Ther. 2006 Feb;5(2):200-8. doi: 10.1158/1535-7163.MCT-05-0420. PMID 16505092
- [Background] Gold DV, Modrak DE, Ying Z, Cardillo TM, Sharkey RM, Goldenberg DM. New MUC1 serum immunoassay differentiates pancreatic cancer from pancreatitis. J Clin Oncol. 2006 Jan 10;24(2):252-8. doi: 10.1200/JCO.2005.02.8282. Epub 2005 Dec 12. PMID 16344318
- [Background] Modrak DE, Cardillo TM, Newsome GA, Goldenberg DM, Gold DV. Synergistic interaction between sphingomyelin and gemcitabine potentiates ceramide-mediated apoptosis in pancreatic cancer. Cancer Res. 2004 Nov 15;64(22):8405-10. doi: 10.1158/0008-5472.CAN-04-2988. PMID 15548711
- [Background] Gold DV, Modrak DE, Schutsky K, Cardillo TM. Combined 90Yttrium-DOTA-labeled PAM4 antibody radioimmunotherapy and gemcitabine radiosensitization for the treatment of a human pancreatic cancer xenograft. Int J Cancer. 2004 Apr 20;109(4):618-26. doi: 10.1002/ijc.20004. PMID 14991585
- [Background] Gold DV, Schutsky K, Modrak D, Cardillo TM. Low-dose radioimmunotherapy ((90)Y-PAM4) combined with gemcitabine for the treatment of experimental pancreatic cancer. Clin Cancer Res. 2003 Sep 1;9(10 Pt 2):3929S-37S. PMID 14506191
- [Background] Modrak DE, Gold DV, Goldenberg DM, Blumenthal RD. Colonic tumor CEA, CSAp and MUC-1 expression following radioimmunotherapy or chemotherapy. Tumour Biol. 2003 Jan-Feb;24(1):32-9. doi: 10.1159/000070658. PMID 12743424
- [Background] Reddy PK, Gold DV, Cardillo TM, Goldenberg DM, Li H, Burton JD. Interferon-gamma upregulates MUC1 expression in haematopoietic and epithelial cancer cell lines, an effect associated with MUC1 mRNA induction. Eur J Cancer. 2003 Feb;39(3):397-404. doi: 10.1016/s0959-8049(02)00700-1. PMID 12565994
- [Background] Cardillo TM, Blumenthal R, Ying Z, Gold DV. Combined gemcitabine and radioimmunotherapy for the treatment of pancreatic cancer. Int J Cancer. 2002 Jan 20;97(3):386-92. doi: 10.1002/ijc.1613. PMID 11774294
- [Background] Cardillo TM, Ying Z, Gold DV. Therapeutic advantage of (90)yttrium- versus (131)iodine-labeled PAM4 antibody in experimental pancreatic cancer. Clin Cancer Res. 2001 Oct;7(10):3186-92. PMID 11595713
- [Background] Gold DV, Cardillo T, Vardi Y, Blumenthal R. Radioimmunotherapy of experimental pancreatic cancer with 131I-labeled monoclonal antibody PAM4. Int J Cancer. 1997 May 16;71(4):660-7. doi: 10.1002/(sici)1097-0215(19970516)71:43.0.co;2-e. PMID 9178823
- [Background] Mariani G, Molea N, Bacciardi D, Boggi U, Fornaciari G, Campani D, Salvadori PA, Giulianotti PC, Mosca F, Gold DV, et al. Initial tumor targeting, biodistribution, and pharmacokinetic evaluation of the monoclonal antibody PAM4 in patients with pancreatic cancer. Cancer Res. 1995 Dec 1;55(23 Suppl):5911s-5915s. PMID 7493369
- [Background] Alisauskus R, Wong GY, Gold DV. Initial studies of monoclonal antibody PAM4 targeting to xenografted orthotopic pancreatic cancer. Cancer Res. 1995 Dec 1;55(23 Suppl):5743s-5748s. PMID 7493339
- [Background] Gold DV, Alisauskas R, Sharkey RM. Targeting of xenografted pancreatic cancer with a new monoclonal antibody, PAM4. Cancer Res. 1995 Mar 1;55(5):1105-10. PMID 7866995
- [Background] Gold DV, Lew K, Maliniak R, Hernandez M, Cardillo T. Characterization of monoclonal antibody PAM4 reactive with a pancreatic cancer mucin. Int J Cancer. 1994 Apr 15;57(2):204-10. doi: 10.1002/ijc.2910570213. PMID 7512537